CLINICAL TRIAL: NCT05963607
Title: RCT of a Weighted Blanket to Reduce Pain in Veterans With Chronic Pain
Acronym: WB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NURP-005-22F; I01CX002591 (NIH)
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Sleep Disturbance
Keywords: chronic pain; sleep; weighted blanket; mood
MeSH Terms: conditions — Chronic Pain; Parasomnias

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with two study arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked to study group to the extent possible (blanket weights are self-evident). Data will be collected online/remotely with no interaction from the study team except for study reminders or technical assistance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heavy blanket (Experimental): Wear heavy blanket overnight for 6 weeks
  Interventions: Other: Weighted blanket
- Light blanket (Active Comparator): Wear light blanket overnight for 6 weeks
  Interventions: Other: Weighted blanket

INTERVENTIONS:
Other: Weighted blanket — A blanket sewn with extra weight in it.

SUMMARY:
Chronic pain is a major health concern for returning Veterans and is associated with decreases in quality of life. In addition, chronic pain is often accompanied by significant disturbance in sleep. Sensory interventions may offer effective, low-cost complementary tools for chronic pain and sleep disturbance in Veterans. Weighted Blankets (WB)- blankets sewn with weighted material inside to provide widespread pressure to the body- are a low-cost wellness product used for anxiety and sleep. WBs have demonstrated large reductions in insomnia, and the investigators have also shown that they can reduce the severity of chronic pain. However, effects and mechanisms of longer WB use have not been examined in individuals with pain and sleep disturbance. The investigators therefore propose a randomized controlled trial examining the effects of WBs on pain and sleep quality in Veterans. the investigators will recruit Veterans with chronic pain and sleep disturbance from the VA San Diego Healthcare System (VASDHS) and VA San Francisco Healthcare System (VASFHS) and randomize 160 Veterans to receive either a light (3-lb; N = 80) or heavy (15-lb; N = 80) blanket. The investigators will remotely collect measures of pain (primary), pain catastrophizing, and pain medication use, as well as sleep disturbance (primary) and sleep efficiency and total sleep time over 6 weeks of overnight home use of the assigned blanket. The investigators will also explore physiological effects of WBs on sleep quality using actigraphy (exploratory) in VASDHS participants. Ecological momentary assessment (EMA) methods will be deployed via smartphone to capture study adherence.

DETAILED DESCRIPTION:
Chronic pain is a major health concern for returning Veterans15 and is associated with decreases in quality of life16, increased opioid use/misuse and self-injury17,18, and significant emotional toll on the patient and medical provider19. The management of pain is a high priority for the Veterans Administration (VA)20 and VA primary care providers21. In addition, chronic pain is highly comorbid with significant disturbance in sleep22, and sleep fragmentation and poor sleep, in turn, are associated with increases in pain sensitivity and pain interference23,24. Decreasing sleep disturbance among Veterans with chronic pain therefore has the potential to greatly reduce pain22, ultimately improving quality of life.

Sensory interventions may offer effective, low-cost complementary tools for chronic pain and sleep disturbance in Veterans. Deep pressure is pleasant and calming25, and reduces acute pain8 and anxiety25 in healthy adults. Weighted Blankets (WB)- blankets sewn with weighted material inside to provide widespread pressure to the body- are a low-cost wellness product used for anxiety and sleep. WBs have demonstrated large reductions in insomnia in individuals with (Cohen's d = 1.9)11 and without12 psychiatric disorders, as well as significant reductions in anxiety and sympathetic arousal26. Tm nl;phe investigators have demonstrated that 1-week of overnight WB use can also reduce chronic pain (severity/interference)27. However, effects and mechanisms of longer WB use have not been examined in individuals with pain and sleep disturbance. The investigators posit that pressure from a WB reduces pain and anxiety while falling asleep and sleeping, decreasing sleep fragmentation and sleep disturbance overnight and, in turn, decreasing pain and pain catastrophizing. The investigators therefore propose a randomized controlled trial examining the effects of WBs on pain and sleep quality in Veterans.

The two objectives of this CSR&D Merit Review are to determine whether in Veterans with musculoskeletal chronic pain and sleep disturbance, a heavy WB versus light (control) blanket will reduce pain impact (severity/interference) and sleep disturbance, and whether improvements in sleep mediate such reductions in pain. The investigators will recruit Veterans with chronic pain and sleep disturbance from the VA San Diego Healthcare System (VASDHS) and VA San Francisco Healthcare System (VASFHS) and randomize 160 Veterans to receive either a light (3-lb; N = 80) or heavy (15-lb; N = 80) blanket. The investigators will collect measures of pain (primary), pain catastrophizing, and pain medication use, as well as sleep disturbance (primary) and sleep efficiency and total sleep time over 6 weeks of overnight use of the assigned blanket. The investigators will also explore physiological effects of WBs on sleep quality using actigraphy (exploratory) in VASDHS participants. Ecological momentary assessment (EMA) methods will be deployed via smartphone to capture study adherence. Our central hypothesis is that although both study arms will be associated with positive clinical outcomes, deeper pressure from the WB will be associated with significantly greater reductions in pain impact and sleep disturbance, with improvements in sleep mediating reductions in pain. The investigators will examine the following aims:

Aim1: Compare the efficacy of a WB versus control blanket on pain in Veterans with musculoskeletal chronic pain and sleep disturbance. Hypothesis 1a: Pain impact (severity and interference) measured by the Pain, Enjoyment of Life, and General Activity (PEG) Scale28 (primary outcome) and pain catastrophizing (Pain Catastrophizing Scale; PCS)29 will show significantly greater improvement in a group of Veterans with chronic pain over 6 weeks from nightly use of a 15-lb versus 3-lb blanket. Hypothesis 1b: Veterans with chronic pain using the 15-lb versus 3-lb blanket will show significantly greater reductions in pain medication use. Exploratory Hypothesis 1c: Pain impact of 15 vs 3-lb blanket will remain higher 12-weeks after randomization.

Aim2: Compare the efficacy of a WB versus control blanket on sleep disturbance in Veterans with musculoskeletal chronic pain and sleep disturbance. Hypothesis 2a: Veterans using the 15-lb versus 3-lb blanket will show significantly greater improvement in sleep disturbance (Insomnia Severity Index; ISI30; primary outcome measure) and sleep efficiency and total sleep time (Daily Sleep Diary31,32) over 6 weeks of use of a 15-lb versus 3-lb blanket. Exploratory Hypothesis 2b: Veterans using the 15-lb versus 3-lb blanket will show increased sleep efficiency and total sleep time (measured by actigraphy) after six weeks of use.

Aim3: Examine the mediation effect of sleep on pain. Hypothesis 3a: Decreases in sleep disturbance (Insomnia Severity Index; ISI30) will mediate reductions in pain impact (PEG28) over the 6-week intervention. Exploratory Hypothesis 3b: Improvements in sleep efficiency (actigraphy) will mediate reductions in PEG pain.

Our expected outcomes are to identify the effects of a WB on chronic pain and sleep disturbance, and the relationship between these clinical factors. The proposed research findings will have a positive impact by providing evidence for effects on chronic pain and sleep disturbance for this novel, accessible and fully remote intervention. Study results will inform both future research and treatment of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

The inclusion/exclusion criteria are designed to be as inclusive as possible and to reflect the heterogeneity of "real-world" Veterans referred to usual care, to maximize generalizability:

* VA-enrolled
* All genders, ages 18 and older
* chronic non-cancer musculoskeletal pain diagnosis on 2 clinical visits for at least 6 months (ICD codes for chronic pain), and a score of 3 on the numerical pain rating scale from 0-10 over the past week
* sleep disturbance measured by a score >= 11 on the ISI.

Exclusion Criteria:

Exclusion criteria: Exclusion criteria include only those factors that contraindicate usual treatment for chronic pain, that prevent the Veteran from benefiting from study treatments, or that may interfere with the mechanisms under study:

* Serious or untreated mental illness (e.g., psychosis; PTSD will not be excluded),
* other psychosocial instability (e.g., homelessness), or
* suicidal/homicidal ideation/prior attempt within the past 3 years by the Mini-International Neuropsychiatric Interview (MINI)19;
* evidence of opioid use disorder by chart review, or a Current Opioid Misuse Measure (COMM20) score of 9 or both;
* major medical conditions or medical counterindications to use of a 15-lb WB (e.g., self-reported or documented current pregnancy;
* claustrophobia;
* spinal cord injury;
* inability to safely lift 15lb);
* obstructive sleep apnea if untreated, OR STOP-BANG score in "high-risk" category; and
* currently sleeping with a special blanket (such as weighted or cooling blanket).
* Those receiving mental health or other pain treatment will be excluded if there are changes to treatment (either therapy or medications) in the 3 months prior to enrollment or anticipated during the 2-month trial (self-report, confirmed as possible in electronic health record).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain impact change | Weeks 0, 2, 4, and 6
  Pain impact (severity and interference) will be measured by the Pain, Enjoyment of Life, and General Activity (PEG) Scale
Sleep disturbance change | Weeks 0, 2, 4, and 6
  Sleep disturbance will be measured by the Insomnia Severity Index (ISI)

SECONDARY OUTCOMES:
Pain catastrophizing | Weeks 0, 2, 4, and 6
  Pain catastrophizing will be measured by the Pain Catastrophizing Scale (PCS).
Pain medication use | Weeks 0, 2, 4, and 6
  Participants will be asked to self report their current pain medication use including prescribed pain medications, dose, and frequency. Prescriptions will be verified with VA electronic health records. Change in pain medications will be quantified as a percent in daily dose from baseline (if multiple pain medications are prescribed, percent change will be averaged across all pain medications). Opioids will be standardized in morphine milligram equivalents.
Daily Sleep Diary | Weeks 0, 2, 4, and 6
  This 12-item scale measures sleep efficiency and total sleep time.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Strigo, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California

IPD SHARING:
Plan to Share IPD: No